CLINICAL TRIAL: NCT00285259
Title: A Phase 2 Clinical Trial to Evaluate the Safety, Immunogenicity, and Clinical Benefit of a CMV Immunotherapeutic Vaccine in Donors and CMV-Seropositive Recipients Undergoing Allogeneic, Matched Hematopoietic Cell Transplant (HCT)
Brief Title: Cytomegalovirus (CMV) Vaccine in Donors and Recipients Undergoing Allogeneic Hematopoietic Cell Transplant (HCT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Vical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CB01-202
Record Dates: First submitted 2006-01-30; First posted 2006-02-01 (Estimated); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Acute Lymphoblastic Leukemia; Chronic Myelogenous Leukemia; Acute Myelogenous Leukemia; Hodgkin's Lymphoma; Non-Hodgkin's Lymphoma; Myelodysplastic Syndrome
Keywords: cytomegalovirus infection; infectious disease; viremia; cytomegalovirus disease; stem cell transplant; allogeneic; bone marrow transplant; hematopoietic cell transplant; Acute Lymphoblastic Leukemia; Chronic Myelogenous Leukemia; Acute Myelogenous Leukemia; Hodgkin's Lymphoma; Non-Hodgkin's Lymphoma; Myelodysplastic Syndrome
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Acute; Hodgkin Disease; Lymphoma, Non-Hodgkin; Myelodysplastic Syndromes; Cytomegalovirus Infections; Communicable Diseases; Viremia | interventions — VCL-CB01 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VCL-CB01 (Experimental)
  Interventions: Biological: VCL-CB01
- Placebo (Placebo Comparator): PBS
  Interventions: Other: Phosphate-buffered Saline (PBS)

INTERVENTIONS:
Biological: VCL-CB01 — 5 mg/mL, Intramuscular (IM.) 3 vaccinations for donors; 1 vaccination pretransplant, up to 3 vaccinations after transplant for recipients
  Arms: VCL-CB01
Other: Phosphate-buffered Saline (PBS) — 1 mL, IM. 3 vaccinations for donors; 1 vaccination pretransplant, up to 3 vaccinations after transplant for recipients
  Arms: Placebo

SUMMARY:
The purpose of this trial is to evaluate a CMV vaccine given to related donor/recipient pairs (donors prior to peripheral blood stem cell donation and CMV-seropositive recipients just before and after transplantation) and CMV-seropositive recipient-only subjects (related or unrelated) to determine incidence rates of CMV infection, disease, and other complications from immunosuppression and/or transplantation. The outcomes for the groups receiving CMV vaccine will be compared to the outcomes for the group that received the placebo vaccine to see if there is a clinical benefit. For this trial, donors and recipients must have matched HLA genotype (matched at 5/6 or 6/6 HLA loci).

DETAILED DESCRIPTION:
This study was run by Vical and the record was transferred to Astellas on 1/8/2013.

Trial will enroll up to 240 subjects (160 recipients and 80 donors). Qualified donors and/or CMV-seropositive recipients (donor/recipient pairs or recipient-only subjects) will be assigned randomly to receive either a CMV vaccine or a placebo vaccine. Donors will receive 3 vaccines prior to donation and recipients will receive 1 vaccine pretransplant and up to three vaccines posttransplant. Recipients will be followed for up to 1 year after transplant to evaluate the safety of the vaccine and to see if there is a clinical benefit in the group that received the CMV vaccine. The incidence rates of CMV infection, disease, and other complications from immunosuppression and/or transplantation will be studied.

ELIGIBILITY:
Inclusion Criteria:

* males and females age 18-65
* 5/6 or 6/6 classic HLA allele-matched donor
* planned GCSF-mobilized peripheral blood stem cell transplant
* CMV-seropositive recipient
* planned transplant with minimal or no T-cell depletion
* Acute Lymphoblastic Leukemia (ALL) in first or second remission; Acute Myeloid Leukemia (AML) in first or second remission; Chronic Myelogenous Leukemia (CML) in first chronic or accelerated phase, or in second chronic phase; Hodgkin's and non-Hodgkin's lymphoma; myelodysplastic syndrome

Exclusion Criteria:

* planned prophylactic cytomegalovirus antiviral therapy
* planned immunosuppression with alemtuzumab (CAMPATH-IH)
* planned prophylactic therapy with CMV immunoglobulin
* autoimmune disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2006-01-31 (Actual); Primary Completion 2009-11-30 (Actual); Study Completion 2010-11-30 (Actual)

PRIMARY OUTCOMES:
Safety of CMV immunotherapeutic vaccine in donors and recipients undergoing HCT | 1 year
occurrence rate of clinically significant CMV viremia in recipients receiving CMV immunotherapeutic vaccine. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Richard T. Kenney, MD, Study Chair — Vical
Locations (22):
- United States (22):
  - Arizona Cancer Center, Tucson, Arizona
  - City of Hope National Medical Center, Duarte, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - University of Kansas Medical Center, Westwood, Kansas
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center # 408, Hackensack, New Jersey
  - Roswell Park Cancer Institute Corporation, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Strong Memorial Hospital, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - North Carolina Baptist Hosptial, Winston-Salem, North Carolina
  - Baylor University Medical Center, Dallas, Texas
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Background] Kharfan-Dabaja MA, Boeckh M, Wilck MB, Langston AA, Chu AH, Wloch MK, Guterwill DF, Smith LR, Rolland AP, Kenney RT. A novel therapeutic cytomegalovirus DNA vaccine in allogeneic haemopoietic stem-cell transplantation: a randomised, double-blind, placebo-controlled, phase 2 trial. Lancet Infect Dis. 2012 Apr;12(4):290-9. doi: 10.1016/S1473-3099(11)70344-9. Epub 2012 Jan 10. PMID 22237175
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website — https://www.clinicaltrials.astellas.com/study/CB01-202/
- See also: Link to plain language summary of the study on Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=25141&tenant=MT_AST_9011